CLINICAL TRIAL: NCT05939544
Title: Impact of Short-term Supplementation with a Milk Fat Globule Membrane-enriched Powdered Ingredient on Cardiometabolic and Cognitive Health Outcomes
Brief Title: Impact of Milk Fat Globule Membrane Supplementation on Heart and Brain Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Dr Oonagh Markey, Principal Investigator, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 10260
Record Dates: First submitted 2023-06-23; First posted 2023-07-11 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Cardiovascular Diseases; Overweight and Obesity; Cognition
Keywords: milk fat globule membrane; milk polar lipids; cholesterol; cardiometabolic risk
MeSH Terms: conditions — Cardiovascular Diseases; Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Milk Fat Globule Membrane-enriched Powdered Ingredient (Experimental): Participants will be provided with pre-weighed, foil sachets containing a ready-to-mix flavoured powdered supplement that is rich in milk fat globule membrane (and associated complex milk lipids). They will be asked to consume two sachets daily (mixed with water) during the 4-week study period. Sachets will be coded to maintain study blinding.
  Interventions: Dietary Supplement: Experimental: Milk Fat Globule Membrane-enriched Powdered Ingredient
- Control (Placebo) Powdered Ingredient (Placebo Comparator): Participants will be provided with pre-weighed, foil sachets containing an energy- and macronutrient-matched ready-to-mix powdered placebo supplement that is devoid of milk fat globule membrane (and associated complex milk lipids). They will be asked to consume two sachets daily (mixed with water) during the 4-week study period. Sachets will be coded to maintain study blinding.
  Interventions: Dietary Supplement: Placebo Comparator: Control (Placebo) Powdered Ingredient

INTERVENTIONS:
Dietary Supplement: Experimental: Milk Fat Globule Membrane-enriched Powdered Ingredient — Milk Fat Globule Membrane-enriched Powdered Ingredient
  Arms: Milk Fat Globule Membrane-enriched Powdered Ingredient
Dietary Supplement: Placebo Comparator: Control (Placebo) Powdered Ingredient — Placebo Comparator: Control (Placebo) Powdered Ingredient
  Arms: Control (Placebo) Powdered Ingredient

SUMMARY:
In a randomised, controlled cross-over manner, this trial aims to determine how short-term daily supplementation with a milk fat globule membrane-enriched ingredient impacts on cardiometabolic health and cognitive outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 - 70 years
* BMI: 25-45 kg/m2
* Recreationally active (> 3 x 30 min moderate exercise per week)
* Understands and is willing and able to comply with all study procedures, including changes to diet
* Fluent in written and spoken English
* Access to, and able to use, the internet/computer/tablet device

Exclusion Criteria:

* Smoking (including vaping)
* Unstable weight history (≥3 kg loss or gain in the previous 3 months) or planning or currently on a weight reduction scheme
* Currently taking part or have participated in another research study in the last two months (e.g., dietary intervention)
* Diagnosed with cardiovascular disease or suffered myocardial infarction/stroke in the past twelve months
* Existing or significant past medical history of any medical condition likely to affect the study outcomes.
* Prescribed medications or supplements likely to interfere with study outcomes or prescribed antibiotics within the last three months
* Use of antidepressant/anti-anxiety medication if it has changed in the last three months or expected to change within the 3-month study period.
* Known allergy or intolerance to study food (lactose intolerance, dairy)
* Being vegan or any other unusual medical history or diet and lifestyle habits or practices that would preclude volunteers from participating in a dietary intervention or metabolic study
* Excessive alcohol consumption: >21 unit/wk
* Pregnancy, seeking to become pregnant or active lactation

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Change-from-baseline in circulating LDL-cholesterol concentrations | 28 days
  Assessed following the collection of fasted blood samples before and after each 28-day study period

SECONDARY OUTCOMES:
Change-from-baseline in circulating lipid and apolipoprotein concentrations (measured using a spectrophotometric assay or high-throughput 1H-NMR metabolomics platform) | 28 days
  Assessed following the collection of fasted blood samples before and after each 28-day study period
Change-from-baseline in particle size of lipoprotein subclasses, and concentrations of particles within each subclass by high-throughput 1H-NMR metabolomics platform | 28 days
  Assessed following the collection of fasted blood samples before and after each 28-day study period
Change-from-baseline in interleukin-6 concentrations (determined by ELISA) | 28 days
  Assessed following the collection of fasted blood samples before and after each 28-day study period
Change-from-baseline in lipopolysaccharide-binding protein concentrations (determined by ELISA) | 28 days
  Assessed following the collection of fasted blood samples before and after each 28-day study period
Change-from-baseline in selected gut-related metabolites (for example, trimethylamine N-oxide concentrations determined by mass spectrometry) | 28 days
  Assessed following the collection of fasted blood samples before and after each 28-day study period
Change-from-baseline in glucose concentrations (determined by spectrophotometric assay) | 28 days
  Assessed following the collection of fasted blood samples before and after each 28-day study period
Change-from-baseline in insulin concentrations (determined by ELISA) | 28 days
  Assessed following the collection of fasted blood samples before and after each 28-day study period
Change-from-baseline in HOMA-IR (calculated as [fasting glucose (mmol/L) × fasting insulin (mIU/L)]/22.5]) | 28 days
  Assessed following assessment of fasting circulating glucose and insulin concentrations before and after each 28-day study period
Change-from-baseline in clinic systolic and diastolic blood pressure (assessed by automated upper arm sphygmomanometer) | 28 days
  Assessed in the fasted state before and after each 28-day study period
Change-from-baseline in arterial stiffness, as assessed by radial pulse wave analysis (using applanation tonometry) | 28 days
  Assessed in the fasted state before and after each 28-day study period
Change-from-baseline in forearm blood flow, as assessed by venous occlusion plethysmography (using applanation tonometry) | 28 days
  Assessed in the fasted state before and after each 28-day study period
Change-from-baseline in cognitive test performance using a neuropsychological seven-test battery which assesses global and domain specific function, as determined by NeurOn software | 28 days
  Assessed before and after each 28-day study period
Change-from-baseline in brain-derived neurotrophic factor concentrations (determined by ELISA) | 28 days
  Assessed in the fasted state before and after each 28-day study period
Change-from-baseline in body mass (kg) using standard equipment. | 28 days
  Assessed in the fasted state before and after each 28-day study period
Change-from-baseline in waist circumference (cm) using standard equipment. | 28 days
  Assessed in the fasted state before and after each 28-day study period
Change-from-baseline in body fat (%) using standard equipment. | 28 days
  Assessed in the fasted state before and after each 28-day study period

CONTACTS AND LOCATIONS:
Locations (1):
- Loughborough University, Loughborough, United Kingdom

IPD SHARING:
Plan to Share IPD: No